CLINICAL TRIAL: NCT01378286
Title: A Randomised Comparative Study to Assess the Efficacy and Tolerability of Blood Schizonticidal Treatments With Artesunate Amodiaquine Winthrop® / Coarsucam (ASAQ) Versus Chloroquine (CQ) for Uncomplicated Plasmodium Vivax Monoinfection Malaria
Brief Title: Efficacy and Tolerability of Artesunate Amodiaquine Versus Chloroquine in the Treatment of Uncomplicated Plasmodium Vivax Malaria
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ARAMF_C_05370; U1111-1120-0233 (Other: UTN)
Record Dates: First submitted 2011-06-20; First posted 2011-06-22 (Estimated); Last update posted 2013-07-18 (Estimated); Status verified 2013-07

CONDITIONS: Malaria
MeSH Terms: conditions — Malaria | interventions — amodiaquine, artesunate drug combination; Chloroquine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- artesunate/amodiaquine (Experimental): artesunate (AS) / amodiaquine (AQ) as fixed dose combination
  1 tablet of AS 25mg/ AQ 67,5mg or AS 50mg/AQ 135mg or AS 100mg/ AQ 270mg or 2 tablets of AS 100mg/ AQ 270mg dose according to bodyweight Once daily 3 days of treatment
  Interventions: Drug: ARTESUNATE + AMODIAQUINE
- chloroquine (Active Comparator): 150mg tablets 25mg/kg in 3 days (10mg/kg on day 1 and 7,5 mg/kg on days 2 and 3) dose according to bodyweight Once daily 3 days of treatment
  Interventions: Drug: Chloroquine

INTERVENTIONS:
Drug: ARTESUNATE + AMODIAQUINE — Pharmaceutical form:
  Route of administration:
  Arms: artesunate/amodiaquine
Drug: Chloroquine — Pharmaceutical form:tablet Route of administration: oral
  Arms: chloroquine

SUMMARY:
Primary Objective:

- To demonstrate the non-inferiority of corrected adequate clinical and parasitological response at Day 28 of Artesunate Amodiaquine (ASAQ) versus chloroquine

Secondary Objectives:

* To assess the non inferiority on the same way as the main criteria:
* at Day 28 before corrected cure rate
* at Day 14 and Day 42 before and after corrected cure rate
* To compare the two groups of treatment in terms of:
* Efficacy:

  * Proportion of aparasitaemic patients at 24, 48 an 72 hours
  * Proportion of afebrile patients at 24, 48 and 72 hours
  * Percentage of gametocyte carriers during follow-up
  * Evolution of the mean of gametocytes during the 42 days of follow-up
  * Evolution of haemoglobin value between Day 0 and Day 7, Day 0 and Day 28
* Clinical and biological tolerability:

  * Proportion of any adverse event
  * Biological safety: haematology (Red blood cells, Haemoglobin, White Blood Cells, neutrophils, platelets), biochemistry (creatinine, transaminases (alanine amino transferase/ALT), bilirubins)
  * ECG (electro encephalogram) (Day 0, Day 3,Day 28) only for patients 10 years old and above

DETAILED DESCRIPTION:
Each patient will be followed for a period of 42 days

ELIGIBILITY:
Inclusion criteria:

* Adults and children over 6 months old and bodyweight > 5 kg
* Able to be treated by oral route
* Axillary temperature ≥ 37,5 C or history of fever during the previous 2 days
* Symptomatic biologically confirmed Plasmodium vivax mono-infection, with parasitemia from 250 to 100000 parasites /µl of blood
* Written informed consent of the patients and for children written informed consent of the parents/legal representative for children. Children able to understand the objectives and the risks of the study will sign an assent form.

Exclusion criteria:

* Known project of leaving the investigator site area during the follow-up period (42 days)
* Hypersensitivity to one of the investigational medicinal products or to any of the excipients
* Intake of an antimalarial treatment in the previous 30 days
* History of hepatic and (or) haematological impairment during treatment with amodiaquine
* Blurred vision suggesting a retinopathy
* Presence of at least one danger sign of malaria
* Pregnant or breast-feeding women
* Women with childbearing potential not willing to use an effective contraceptive method(s) for the duration of the study
* Known severe concomitant or underlying disease

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Min Age: 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 380 (Actual)
Dates: Start 2012-01; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Assessment of clinical and parasitological efficacy based on temperature and parasitemia after Polymerase chain reaction (PCR) correction | 28 days

SECONDARY OUTCOMES:
Assessment of clinical and parasitological efficacy based on temperature and parasitemia before and after PCR correction at D14 and D42 and before PCR correction at D28 | up to a maximum of 42 days
Number of patients without parasite | up to a maximum of 42 days
Number of patients without fever | up to a maximum of 42 days
Number of patients with gametocytes | up to a maximum of 42 days
Change from baseline in Haemoglobin levels | Day 7, Day 28
Incidence and severity of adverse events collected | up to a maximum of 42 days
ECG (QTc) changes in patients group aged >= 10 years from baseline | Day 3, Day 28
Assessment of biological tolerability (bilirubin, ALAT, Creatinine, Leukocytes, Neutrophils and platelets count) from baseline | up to a maximum of 42 days

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (1):
- Administrative office, São Paulo, Brazil

REFERENCES:
- [Derived] Siqueira AM, Alencar AC, Melo GC, Magalhaes BL, Machado K, Alencar Filho AC, Kuehn A, Marques MM, Manso MC, Felger I, Vieira JL, Lameyre V, Daniel-Ribeiro CT, Lacerda MV. Fixed-Dose Artesunate-Amodiaquine Combination vs Chloroquine for Treatment of Uncomplicated Blood Stage P. vivax Infection in the Brazilian Amazon: An Open-Label Randomized, Controlled Trial. Clin Infect Dis. 2017 Jan 15;64(2):166-174. doi: 10.1093/cid/ciw706. Epub 2016 Oct 20. PMID 27988484